CLINICAL TRIAL: NCT04866537
Title: Evaluation of the Diagnostic Performance of Specialized Fetal Cardiac Ultrasound in the CPDPN - Arc Alpin Network From 2015 to 2019 Descriptive, Retrospective, Single-center Study Over 5 Years.
Brief Title: Evaluation of the Diagnostic Performance of Specialized Fetal Cardiac Ultrasound in the CPDPN - Arc Alpin Network
Acronym: Qualicard
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A01842-37
Record Dates: First submitted 2021-04-28; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Heart Defects, Congenital; Ultrasonography, Prenatal
Keywords: Heart Defects, Congenital / diagnostic imaging
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women who received a fetal heart ultrasound between 2015 and 2019.: Pregnant women who received a fetal heart ultrasound between 2015 and 2019.

SUMMARY:
To evaluate the diagnostic performance of antenatal echocardiography with regard to the main diagnosis of heart disease made by cardio-pediatricians at the couple-child hospital in Grenoble according to the ACC-CHD classification, in pregnant women who have had a fetal heart ultrasound between 2015 and 2019.

*ACC-CHD : Anatomic and Clinical Classification of Congenital Heart Defects

DETAILED DESCRIPTION:
This work is in line with the desire of the Pluridisciplinary Center for Pre-Natal Diagnosis (CPDPN) of the Arc Alpin network, to assess their professional practices regarding the prenatal diagnosis of heart disease over the last five years from 2015 to 2019, and so identify areas for improving their care.

Within the Arc-Alpin network, pregnant women for whom an abnormality is detected in the fetus during the screening ultrasound, then benefit from a diagnostic ultrasound, to confirm the detected abnormality. Then, the patient's file will be studied within the CPDPN of the Alpine Arc, and the patient will then be referred to a doctor specializing in the diagnosed fetal pathology. The latter will prescribe additional examinations to characterize as much as possible the diagnosed pathology, in order to develop a course of action to be taken, and to establish a prognosis for this fetus (specialized ultrasound, MRI, amniocentesis, etc.)

As part of the diagnosis of fetal heart disease, the woman will be referred to cardio-pediatricians at the Couple Enfant Hospital in Grenoble, who will perform a so-called specialized 2nd line ultrasound in order to clarify the diagnosis, to develop a course of action to take, and establish a prognosis for this unborn child.

We therefore want to study the diagnostic performance of specialized 2nd line fetal cardiac ultrasound in the CPDPN network of the Alpin Arc, by comparing the diagnosis established following the 2nd line fetal echocardiography with the reference examination (test of reference) which is the postnatal cardiac ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who have had a fetal heart ultrasound performed by a cardiac pediatrician at the Hopital Couple Enfant in Grenoble between 2015 and 2019.

Exclusion Criteria:

- No

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Pregnant women who have had a fetal heart ultrasound performed by a cardiac pediatrician at the Hopital Couple Enfant in Grenoble between 2015 and 2019.
Sampling Method: Probability Sample
Enrollment: 679 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the diagnostic performance of antenatal echocardiography with regard to the main diagnosis of heart disease made by cardio-pediatricians at the Grenoble couple-child hospital according to the ACC-CHD classification. | 5 years
  Sensitivity of fetal echocardiography to the primary diagnosis of heart disease made by cardio-pediatricians.

SECONDARY OUTCOMES:
Evaluation of the diagnostic performance of antenatal echocardiography with regard to the main diagnosis of heart disease made by cardio-pediatricians in each pathology sub-category of the ACC-CHD classification. | 5 years
  Sensitivity of fetal cardiac ultrasound to the main heart disease diagnosis made by cardio-pediatricians in each pathology subcategory of the ACC-CHD classification.
Evaluation of the diagnostic performance of antenatal echocardiography with regard to secondary diagnoses of heart disease made by cardio-pediatricians. | 5 years
  Sensitivity of fetal echocardiography to secondary heart disease diagnosis made by cardio-pediatricians in each pathology subgroup.

CONTACTS AND LOCATIONS:
Overall Officials: Eline DURAND, Principal Investigator — CHU GRENOBLE ALPES - IFPS - Département de Maïeutique
Locations (1):
- Centre Hospitalier Universitaire GRENOBLE ALPES, Grenoble, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: Undecided